CLINICAL TRIAL: NCT02540655
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Single-Center Study to Evaluate the Safety and Efficacy of Stemchymal® Infusion for the Treatment of Polyglutamine Spinocerebellar Ataxia
Brief Title: Efficacy and Safety Study of Stemchymal® in Polyglutamine Spinocerebellar Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steminent Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IB02
Record Dates: First submitted 2015-08-26; First posted 2015-09-04 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Cerebellar Ataxia
Keywords: Stem Cells; Adult Stem Cells; Spinocerebellar Ataxia; Steminent
MeSH Terms: conditions — Cerebellar Ataxia; Spinocerebellar Ataxias | interventions — Excipients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stemchymal® (Experimental): Infusion of Stemchymal®
  Interventions: Biological: Stemchymal®
- Vehicle (Placebo Comparator): Infusion of excipients
  Interventions: Procedure: Excipients

INTERVENTIONS:
Biological: Stemchymal® — Patients will receive Stemchymal® through intravenous infusion
  Arms: Stemchymal®
Procedure: Excipients — Patients will receive excipients through intravenous infusion
  Arms: Vehicle

SUMMARY:
The purpose of the clinical trial is to study the therapeutic efficacy and safety of Stemchymal® infusions for polyglutamine spinocerebellar ataxia treatment by a randomized, double-blind, placebo-controlled study design. Eligible subjects will receive Stemchymal® through intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are with genotypically confirmed spinocerebellar ataxia type 2 or spinocerebellar ataxia type 3.
2. Subjects' baseline SARA score are in the range of 8 to15.
3. Subjects are between 20 and 70 years of age.
4. Subjects who had signed informed consent.

Exclusion Criteria:

1. Subjects had been enrolled in any kind of cell therapy within six months prior to screening visit.
2. Females with a positive pregnancy test result.
3. Subjects who had had severe vital organ disease as diagnosed, including but not limited to cardiac (ex. heart failure), liver (ex. acute hepatic failure or chronic liver cirrhosis), lung (ex. respiratory failure) and renal (ex. hemodialysis or peritoneal dialysis) insufficiency, within six months prior to screening visit.
4. Subjects with immunological disorders (ex. Systemic lupus erythematosus), within six months prior to screening visit.
5. Subjects with other neurological disorders (ex. Alzheimer's disease), within six months prior to screening visit.
6. Subjects who had received chemotherapy/radiotherapy within five years prior to screening visit.
7. Subjects with any history of malignancy tumors.
8. Subjects with a history of hypersensitivity/allergy to penicillin.
9. Subjects with dementia or other psychiatric illnesses, including but not limited to disabling depression, bipolar disorder, and schizophrenia.
10. Subjects with Beck Depression Inventory Second Edition (BDI-II) score over 20 points.
11. Subjects with unstable illnesses or contraindication for this clinical trial according to PI's judgment.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-09; Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
To assess the changes from the baseline to all visits on Scale for the Assessment and Rating of Ataxia (SARA) score. | 14 months

SECONDARY OUTCOMES:
To assess the safety by incidence of adverse events, changes of vital signs, blood biochemistry tests, complete blood count, immunoactivity assay, urinalysis and magnetic resonance imaging (MRI). | 14 months
To assess the changes from the baseline to all visits on SCA functional index (SCAFI) | 14 months
To assess the changes from the baseline to all visits on sensory organization test (SOT) | 14 months
  Balance test
To assess the changes from the baseline to all visits on inventory of non-ataxia signs (INAS) | 14 months
To assess the changes from the baseline to all visits on clinical global impression (CGI) | 14 months
To assess the changes from the baseline to all visits on patient global impression of improvement (PGI-I) | 14 months

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan